CLINICAL TRIAL: NCT03455972
Title: Study of T Cells Targeting CD19/BCMA (CART-19/BCMA) for High Risk Multiple Myeloma Followed With Auto-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: myeloma-03
Record Dates: First submitted 2018-02-19; First posted 2018-03-07 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2020-12

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — Immunomodulating Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 and anti-BCMA CAR (Experimental): Participants will get auto-HSCT. Hematopoietic reconstitution after auto-HSCT, participants will get the anti-CD19 CAR T cells (on d0) and anti-BCMA CAR T cells as split-dose (40% on d1 and 60% on d2)
  Interventions: Biological: anti-CD19 and anti-BCMA CAR; Drug: Immunomodulatory drugs

INTERVENTIONS:
Biological: anti-CD19 and anti-BCMA CAR — Participants will get auto-HSCT. Hematopoietic reconstitution after auto-HSCT, participants will get the anti-CD19 CAR T cells (1×10e+7/kg on d0) and anti-BCMA CAR T cells as split-dose (total 5×10e+7/kg, 40% on d1 and 60% on d2)
Drug: Immunomodulatory drugs — Maintenance therapy
  Other Names: IMiDs

SUMMARY:
CART therapy has showed good safety and efficacy in treatment of lymphoma and acute lymphoblastic leukemia. Researchers want to see if this helps people with high risk multiple myeloma after auto-HSCT.To test the safety and efficacy of giving targeting CD19 and BCMA T cells in treating high risk multiple myeloma followed with auto-HSCT.

DETAILED DESCRIPTION:
Adults ages 18-75 with high risk Multiple Myelomas (R-ISS III stage or with extramedullary infiltration or with del(17p), t(4;14), t(14;16), t(14;20), 1q21+ or disease progression during treatment).

Design:

Participants may be screened with:

Medical history Physical exam Blood and urine tests Heart tests Bone marrow sample Multiple scans and X-rays Participants will have apheresis. Blood is removed through a needle in an arm. T cells are removed. The rest of the blood is returned through a needle in the other arm.

The cells will be changed in a laboratory. Participants will get auto-HSCT. Hematopoietic reconstitution after auto-HSCT, participants will get the T cells through the IV within 3 days. Maintenance therapy with IMiDs was received after combined CAR T infusion.

After this, participants will stay in the hospital for at least 9 days and stay nearby for 2 weeks. Then they will have blood tests and see a doctor.

Participants will visit the clinic 1, 2, 3, 6, 9 and 12 months after the infusion, then every 3 months until disease progression. A bone marrow sample will be taken at the 3-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients eligible for auto-HSCT.
* High risk multiple myeloma (R-ISS III stage or with extramedullary infiltration or with del(17p), t(4;14), t(14;16), t(14;20), 1q21+ or disease progression during treatment).
* Expected survival ≥ 3 months.
* Creatinine < 2.0 mg/dl.
* Blood coagulation function: PT and APTT <2x normal.
* Arterial blood oxygen saturation>92%.
* ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal
* Karnofsky scores ≥ 60 and ECOG score≤2.
* Adequate venous access for apheresis, and no other contraindications for leukapheresis.
* Patients should not take immunotherapy in three months prior to CART cells infusion.
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* History of myocardial infarction and severe arrhythmia in half a year.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Patients with fever of unknown origin (T>38℃).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Approximately 3 years
  Proportion of subjects with adverse events overall and by severity grade
PFS | Minimum of 2 years after first induction
  Is defined as time from first induction date to first documentation of PD, or death due to any cause, whichever occurs first.
OS | Minimum of 2 years after first induction
  Is defined as time from first induction date to time of death due to any cause

SECONDARY OUTCOMES:
Duration of best response | Minimum of 2 years
  According to IMWG response criteria at the end of the research.
MRD negative conversion ratio and persistence | Minimum of 2 years
  MRD negative by flow cytometry
Proportion of subjects who achieved Complete Response (CR) Rate | Minimum of 2 years
  Percentage of subjects who achieved CR or stringent CR according to IMWG Uniform Response Criteria for Multiple Myeloma
Pharmacokinetics - Cmax | Approximately 2.5 years after first CAR infused
  Maximum transgene level
Pharmacokinetics - Tmax | Approximately 2.5 years after first CAR infused
  Time to peak transgene level
Pharmacokinetics - AUC | Approximately 2.5 years after first CAR infused
  Area under the curve of the transgene level
Duration of persistence of CAR T cells in the blood | Approximately 2.5 years after first CAR infused
  Duration of persistence of CAR T cells in the blood

CONTACTS AND LOCATIONS:
Overall Officials: depei wu, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China